CLINICAL TRIAL: NCT04354649
Title: A Study to Evaluate the Efficacy and Safety Hydroxychloroquine in Immune Related Arthritis or Arthralgias
Brief Title: Immune-Mediated Pathophysiology And Clinical Triage Program
Acronym: IMPACT 2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIT-0011
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Arthritis; Arthralgia
MeSH Terms: conditions — Arthritis; Arthralgia | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine, plus prednisone (Experimental): Hydroxychloroquine 5mg/kg PO daily, plus prednisone starting at 20 mg PO daily for 8 weeks tapering dose.
  Interventions: Drug: Hydroxychloroquine
- Hydroxychloroquine-matching placebo, plus prednisone (Placebo Comparator): Matching placebo daily, plus prednisone starting at 20 mg PO daily for 8 weeks tapering dose.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 5mg/kg PO daily
  Arms: Hydroxychloroquine, plus prednisone
Other: Placebo — Hydroxychloroquine-matching placebo
  Arms: Hydroxychloroquine-matching placebo, plus prednisone

SUMMARY:
Many people develop joint pain, stiffness and swelling due to their cancer treatment that targets the immune system. The severity of symptoms ranges from mild to debilitating and sometimes requires delaying or stopping cancer treatment.

The usual plan is to discontinue cancer treatment and give relatively high doses of a medication called prednisone (a steroid, which is an anti-inflammatory medication which may suppress the immune system) with a gradual lowering of the dose over several weeks. While this can be effective, prednisone can cause a number of side effects, and it is not known if this is the best or safest treatment.

Hydroxychloroquine is a medication that is often used to treat inflammatory joint pain, such as rheumatoid arthritis, has relatively few side effects when compared to prednisone, and may be effective at treating this condition.

The purpose of this study is to find out whether it is better to receive hydroxychloroquine and prednisone, or prednisone alone for joint pain. To do this, some participants will get hydroxychloroquine and some will receive a placebo (a substance that looks like the study drug but does not have any active or medicinal ingredients). A placebo is used to make the results of the study more reliable.

This is a double-blinded study, which means that neither participants nor the study doctor or study staff will know which group participants are allocated. After 12 weeks of study treatment, the blind will be opened and participants will be informed which treatment was given.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age, or older;
2. Patients must be capable of providing consent to enrolment and treatment.
3. Patients with a performance status of ECOG 0-2 will be eligible for enrolment (see appendix A).
4. Patients with histologically confirmed cancer receiving anti-PD1 or anti-PDL1 monoclonal antibody ICI therapy, either alone or in combination with anti-CTLA4 monoclonal antibody ICI therapy who develop CTCAEv5.0 grade ≥2 arthritis or arthralgia that has developed on, or after, ICI therapy and is felt to be treatment related (irAA).
5. Adequate hepatic and renal function defined by the following laboratory parameters:

   * AST and ALT and alkaline phosphatase ≤ 2.5x ULN,
   * Total bilirubin ≤ 1.5x ULN,
   * Serum creatinine ≤ upper limit of institutional normal OR calculated creatinine clearance of ≥ 60 mL/min using the Cockcroft-Gault formula.
6. Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.
7. Patients of childbearing / reproductive potential should use highly effective birth control methods, during the study treatment period and for a period of 3 months after the last dose of study drug. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly. These may include: hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy and tubal ligation. Double-barrier methods may be acceptable in circumstances when highly effective methods cannot be implemented (e.g. male condom with diaphragm, male condom with cervical cap). Note: Contraceptive requirements for the oncology regiments will apply, if they are more stringent than those for this trial. Abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
8. Female patients who are breast-feeding should discontinue nursing prior to the first dose of study treatment and until 3 months after the last dose of study drug.
9. Male patients should agree to not donate sperm during the study and for a period of at least 3 months after last dose of study drug.
10. Absence of any condition hampering compliance with the study protocol and follow- up schedule; those conditions should be discussed with the patient before registration in the trial.

Exclusion Criteria:

1. History of inflammatory arthritis, including, but not limited to: Rheumatoid arthritis, systemic lupus erythematosus, Sjogren's syndrome, Ankylosing spondylitis or other chronic inflammatory arthritis. Note: Patients with a known history of stable osteoarthritis will not be excluded.
2. Patients with an indication for systemic immunosuppressive medications or corticosteroids. Patients with CTCAEv5.0 grade ≥2 irAE's other than irIAA (ie. colitis, pneumonitis, rash, etc) are not eligible for trial, with the exception of endocrinopathies that are being treated with hormone replacement alone and not systemic immunosuppressive medications or corticosteroids.
3. Patients weighing < 40 kg.
4. Patients with G6PD deficiency, porphyria or psoriasis.
5. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
6. Prolonged corrected QT interval or concurrent medications that prolong QT interval.
7. Diagnosis of immunodeficiency.
8. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
9. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (CTCAEv5.0 Grade ≥ 3).
10. Other severe acute or chronic medical conditions including inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Recurrence of grade ≥2 Immune-Related Arthritis or Arthralgia | Through study completion, an average of 1 year
  Recurrence will be defined as the development of grade ≥2 irAA in a participant whose symptoms initially improved to grade ≤1.
  Symptoms will be investigator assessed and graded according to CTCAEv5.0.

SECONDARY OUTCOMES:
Total Steroid Usage | Through study completion, an average of 1 year
  The total cumulative dose of prednisone measured in mg used by the participant. If corticosteroids other than prednisone are used, their equivalent dosage in mg of prednisone will be calculated and used for this analysis.
Development of immune related adverse events (irAE's) other than irAA | Through study completion, an average of 1 year
  Defined as the emergence of adverse events that were not present at study baseline that are deemed by the investigator to be related to prior use of immune checkpoint inhibitors. Causality will be investigator assessed and graded according to CTCAEv5.0.
Adverse Event | Through study completion, an average of 1 year
  The emergence of new or worsening baseline symptoms, physical findings, or laboratory/imaging abnormalities. Causality to study treatment, immune checkpoint inhibitors, or underlying disease status will be investigator assessed and graded according to CTCAEv5.0.
Re-initiation of immune checkpoint inhibitor therapy | Through study completion, an average of 1 year
  The proportion of participants in each study arm that are re-treated with an immune checkpoint inhibitor.
Response to standard of care treatments after Week 13 Day 1. | From Week 13 Day 1 to Week 52.
  Participants that still have active irAA symptoms of CTCAEv5.0 grade ≥1 after unblinding at Week 13 Day 1 visit who have a change in irAA therapy.
Progression free survival | Upon completion of follow-up period, an average of 3 years after intervention
  The time elapsed between randomization and tumor progression (radiographically or clinically) or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kolinsky, Principal Investigator — AHS-CCI
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada